CLINICAL TRIAL: NCT06764069
Title: Early Feasibility Study to Evaluate an Intravascular Blood Continuous Glucose Sensor in Adults with Diabetes Mellitus
Brief Title: Feasibility Study to Evaluate an Intravascular Blood Continuous Glucose Sensor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Glucotrack (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-001
Record Dates: First submitted 2024-12-13; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; CBGM; CGM; type 2 diabetes; type 1 diabetes; diabetes mellitus, insulin dependent
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Each Participant will be wearing a single investigational sensor.
Masking Description: The participants will not have access to the glucose data from the investigational device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Glucotrack Sensor Lead (Experimental): One Glucotrack Sensor Lead will be inserted per Participant.
  Interventions: Device: Sensor Lead

INTERVENTIONS:
Device: Sensor Lead — The Glucotrack Sensor Lead will be inserted into the subclavian vein, using a Seldinger technique, where it will continuously measure blood glucose levels.

SUMMARY:
The goal of this early first in man clinical trial is to evaluate the safety of an implantable continuous blood glucose monitoring system in participants with Diabetes Mellitus. Safety will be assessed by looking at the absence of procedure or device related adverse events. Additionally, the surgical procedure and device performance will be evaluated.

Key Research Questions:

1. Were there any adverse events associated with the insertion of the Sensor Lead?
2. Did Participants experience any device-related adverse events from the Sensor Lead insertion through the 96-hour observation period and subsequent removal of the Sensor Lead?
3. How effectively did the device capture data during the 96-hour wear period?

DETAILED DESCRIPTION:
Eligible Participants will be inserted with the Sensor Lead of the investigational continuous blood glucose monitoring device and stay in the hospital for a 96-hour observation period.

Glucose measurements, medications and food will be tracked throughout the 96-hour Observation period.

Two 3-hour frequent sample tests (sampling every 15-min for glucose measurement) will occur during the 96-hour Observation period.

After approximately 96-hours is complete the participant will have the Sensor Lead removed and will be discharged after an hour observation post removal. A final follow-up visit will occur approximately 1-week post sensor removal to check on the removal site and formally exit that participant from the study.

All safety events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 to 75 years old inclusive
2. Generally, in good health, as determined by the investigator
3. Clinical diagnosis or type 1 or type 2 diabetes as determined via medical records or source documentation by an individual qualified to make a medical diagnosis
4. Intensive Insulin Therapy - 3 plus injections/day (MDI) or Continuous Subcutaneous Insulin Infusion (CSII)
5. HbA1c <9.0 % in the last 3 months.
6. Study subject has adequate venous access as assessed by investigator or appropriate staff.
7. Willing to comply with study procedures and be admitted to hospital for up to 5 days.
8. Willing to perform up to 7 blood glucose (fingerstick) measurements a day using provided blood glucose meters and strips
9. Willing to wear subcutaneous continuous wear glucose sensor for the duration of the study
10. Willing to always carry study provided Android Phone during study
11. Access to internet for required periodic uploads of study device data
12. BMI in the range 18-35 kg/m2
13. Has the ability to understand and comply with protocol procedures and to provide informed consent (i.e., proficient in both verbal and written communication in English or from a translator (Portuguese to English).

Exclusion Criteria:

1. Currently taking Acetaminophen and unable to switch to another anti-inflammatory or pain reliever
2. Currently being treated with an anticoagulation agent
3. History of Deep Vein Thrombosis (DVT), Pulmonary Embolism (PE), or blood clotting disorder that in the opinion of the Investigator would compromise safety of the study subject.
4. Currently using one of the following non-insulin glucose-lowering agent, SGLT2 and Insulin Secretagogues
5. Female study subject of childbearing potential and has a positive pregnancy screening test
6. Female study subject of childbearing potential who is planning to become pregnant or not using adequate method of contraception deemed reliable by Investigator
7. 1 of more episodes of hypoglycemia or diabetic ketoacidosis (DKA) in the last 6 months requiring care in a medical facility or assistance from another individual to treat.
8. Study subject has a hematocrit (Hct) lower than the normal reference range
9. Known cardiovascular disease considered to be clinically relevant by the investigator
10. Currently undergoing treatment with:

    * Systemic oral or intravenous corticosteroids (current or within the last 8 weeks from screening),
    * Thyroid hormones, unless use has been stable during the past 3 months
11. Significant history of any of the following, that in the opinion of the investigator would compromise safety or successful study participation:

    * Alcoholism
    * Drug abuse
12. Significant acute or chronic illness, that in the opinion of the investigator might interfere with safety or integrity of study results
13. Current participation in another clinical drug or device study
14. Study subject may not be on the research staff of those performing this study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-02-04 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: study device safety as evidence by absence of serious procedure or device related adverse event(s). | From enrollment through 7-days (+/-3 days) post Sensor Lead removal.
  No procedure or device related serious adverse events from implant through the 7 days post-explant appointment.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração (InCor) |, São Paulo, Brazil, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Participants will be identified by a participant ID only. Data that may be provided includes demographic data, as well as glucose results from the investigational and supporting commercial devices.
Supporting Information: CSR, Analytic Code
Time Frame: 6 months post study to support publication(s)
Access Criteria: Statisticians, medical writers. They may be able to access through a direct share site and/or the report may be provided to them.